CLINICAL TRIAL: NCT04755777
Title: Provider Perspectives on Beta-lactam Therapeutic Drug Monitoring Programs in the Critically Ill: a Multicenter Mixed-methods Study
Brief Title: Provider Perspectives on Beta-lactam Therapeutic Drug Monitoring Programs in the Critically Ill
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin Barreto, Principal Investigator, Mayo Clinic
Other Study IDs: 20-007528
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sepsis; Critical Illness
Keywords: pharmacokinetics; therapeutic drug monitoring; mixed methods; implementation science; beta-lactam antibiotic
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to characterize various healthcare practitioners' perspectives on implementation of beta-lactam therapeutic drug monitoring in critical care practice.

ELIGIBILITY:
Inclusion Criteria:

* Providers involved with beta-lactam TDM for critically ill patients

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be obtained from ICU clinicians at three hospitals with distinct beta-lactam dosing and monitoring practices: Royal Brisbane and Women's Hospital in Queensland Australia, University of Florida Health Shands Hospital, Gainesville, Florida, United States, and the Mayo Clinic Hospital in Rochester, Minnesota, United States. The sampling frame will include key clinician stakeholders likely to be involved with beta-lactam TDM in the intensive care unit (i.e., pharmacists, intensivists, infectious diseases experts, medical/surgical trainees, and advanced practice providers).
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of drug level testing recommended | Baseline
  Indication of how many critically ill patients treated with beta-lactams should receive TDM.
Nature of drug level testing recommended | Baseline
  Indication of which types of critically ill patients treated with beta-lactams should receive TDM

SECONDARY OUTCOMES:
Determinants of beta-lactam TDM implementation | Baseline
  List of factors associated with successful beta-lactam TDM implementation

CONTACTS AND LOCATIONS:
Overall Officials: Erin Barreto, Pharm. D.,R.Ph., Principal Investigator — Mayo Clinic
Locations (3):
- United States (2):
  - UF Health Shands, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

REFERENCES:
- [Background] Ausman S, Boehmer K, et al. Open Forum Infectious Diseases. 2022;9(Supplement 2):ofac492.034.
- [Derived] Barreto EF, Chitre PN, Pine KH, Shepel KK, Rule AD, Alshaer MH, Abdul Aziz MH, Roberts JA, Scheetz MH, Ausman SE, Moreland-Head LN, Rivera CG, Jannetto PJ, Mara KC, Boehmer KR. Why is the Implementation of Beta-Lactam Therapeutic Drug Monitoring for the Critically Ill Falling Short? A Multicenter Mixed-Methods Study. Ther Drug Monit. 2023 Aug 1;45(4):508-518. doi: 10.1097/FTD.0000000000001059. Epub 2023 Mar 21. PMID 37076424
- [Derived] Barreto EF, Rule AD, Alshaer MH, Roberts JA, Abdul Aziz MH, Scheetz MH, Mara KC, Jannetto PJ, Gajic O, O'Horo JC, Boehmer KR. Provider perspectives on beta-lactam therapeutic drug monitoring programs in the critically ill: a protocol for a multicenter mixed-methods study. Implement Sci Commun. 2021 Mar 24;2(1):34. doi: 10.1186/s43058-021-00134-9. PMID 33762025
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials